CLINICAL TRIAL: NCT06482034
Title: Effect of N-acetyl Cysteine and Zinc in Management of Head and Neck Cancer Radiotherapy Induced Oral Mucositis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Nadia Hamdy Ibrahim Mohamed Aref, B.D.S, M.S, Master Degree of Oral Medicine & Periodontology, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: M02040230M
Record Dates: First submitted 2024-06-03; First posted 2024-07-01 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-06

CONDITIONS: Radiation-Induced Mucositis
MeSH Terms: interventions — Acetylcysteine; Zinc Sulfate

STUDY DESIGN:
Intervention Model Description: The study is a randomized, controlled, interventional clinical trial conducted at Mansoura University Oncology Hospital. Fifty head and neck cancer patients receiving radiotherapy will be randomized into five groups of ten each. Group I will receive N-acetylcysteine (NAC) sachets (600mg) twice daily, Group II will receive zinc sulfate capsules (25mg) thrice daily, Group III will receive both NAC and zinc sulfate, and Group IV will receive NAC and zinc sulfate after mucositis onset. Group V, the control group, will receive standard care with normal saline mouthwash. The study aims to evaluate the efficacy of NAC, zinc sulfate, and their combination in treating radiotherapy-induced oral mucositis. Mucositis severity will be assessed using the WHO criteria for grading oral mucositis. Patients' consent and ethical approval will be obtained.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Group 1 (Experimental): Intervention Type: Drug Intervention Name: N-acetylcysteine (NAC) Other Intervention Names: NAC Intervention Description: Patients will receive N-acetylcysteine sachets (600mg) twice daily. They will dissolve the NAC sachet in a cup of water, gargle for 60 seconds, and swallow it. The treatment will start 3 days before the beginning of radiotherapy and continue for 2 weeks after the completion of the radiotherapy schedule.
  Interventions: Drug: N-acetyl cysteine
- Group2 (Experimental): Arm 2 Intervention Type: Drug Intervention Name: Zinc sulfate Other Intervention Names: Zinc Intervention Description: Patients will receive zinc sulfate capsules (25mg) thrice daily at 8-hour intervals. The treatment will start 3 days before the beginning of radiotherapy and continue for 2 weeks after the completion of the radiotherapy schedule.
  Interventions: Drug: Zinc sulfate
- Group 3 (Experimental): Arm 3 Intervention Type: Combination Product Intervention Name: N-acetylcysteine (NAC) and zinc sulfate Other Intervention Names: NAC and Zinc Intervention Description: Patients will receive N-acetylcysteine sachets (600mg) twice daily and zinc sulfate capsules (25mg) thrice daily. They will dissolve the NAC sachet in a cup of water, gargle for 60 seconds, and swallow it. The treatment will start 3 days before the beginning of radiotherapy and continue for 2 weeks after the completion of the radiotherapy schedule.
  Interventions: Drug: N-acetyl cysteine; Drug: Zinc sulfate
- Group 4 (Experimental): Intervention Type: Combination Product Intervention Name: N-acetylcysteine (NAC) and zinc sulfate after mucositis onset Other Intervention Names: NAC and Zinc post-mucositis Intervention Description: Patients who already began their radiotherapy and developed oral mucositis will receive N-acetylcysteine sachets (600mg) twice daily and zinc sulfate capsules (25mg) thrice daily. They will dissolve the NAC sachet in a cup of water, gargle for 60 seconds, and swallow it. The treatment will continue for 2 weeks after the completion of the radiotherapy schedule.
  Interventions: Drug: N-acetyl cysteine; Drug: Zinc sulfate
- Group 5 (Active Comparator): Intervention Type: Other Intervention Name: Standard care (normal saline mouthwash) Other Intervention Names: Saline mouthwash Intervention Description: Patients will receive the institutional standard care, which is a normal saline mouthwash. The treatment will start 3 days before the beginning of radiotherapy and continue for 2 weeks after the completion of the radiotherapy schedule. Patients who develop any grade of oral mucositis will be treated according to the institutional standard treatment protocol.
  Interventions: Drug: saline mouth wash

INTERVENTIONS:
Drug: N-acetyl cysteine — N-acetyl cysteine sachets
  Arms: Group 1; Group 3; Group 4
Drug: Zinc sulfate — zinc sulfate capsules
  Arms: Group 3; Group 4; Group2
Drug: saline mouth wash — saline mouth wash
  Arms: Group 5

SUMMARY:
The majority of individuals diagnosed with head and neck cancer, who undergo radiotherapy or concurrent Chemoradiotherapy, experience oral mucositis. Our research focuses on investigating the preventive and therapeutic impact of N-acetylcysteine and zinc in managing radiotherapy-induced oral mucositis.

DETAILED DESCRIPTION:
almost all head and neck cancer patients who to receive radiotherapy or concurrent chemotherapy suffer from oral mucositis. Oral mucositis (OM) is associated with pain, difficulty in eating, dysphagia, and the need for enteral or parenteral nutrition, increased opioid consumption or even interruptions to cancer therapy. In immunosuppressed patients, OM is associated with bacteremia, increased inpatient hospitalization duration and higher 100-day mortality.

Treatments to manage cancer, such as radiotherapy, generates reactive oxygen species (ROS) that target neoplastic cell DNA resulting in cell damage and death. ROS from these therapies also indiscriminately target healthy non-neoplastic DNA.

Zinc carries out its antioxidant function in two ways: Reducing the concentration of oxidant agents and protecting structures and macromolecules suffer from oxidant agent.

N-acetylcysteine is an aminothiol and precursor to glutathione (GSH), glutathione in its reduced form is the most powerful intracellular antioxidant, thereby protecting against radiation-induced free radical damage.

our study is A randomized, controlled, parallel clinical trial that will be applied at Clinical Oncology and Nuclear Medicine Center at Mansoura University Hospital to investigate the prophylactic and therapeutic effect of N-acetylcysteine and zinc on radiotherapy induced oral mucositis in Head and Neck cancer patients.

ELIGIBILITY:
Eligibility Criteria

Inclusion Criteria:

* Patients aged 18 years or older.
* Patients diagnosed with head and neck cancer.
* Patients are recommended for treatment with radiotherapy with a minimum dose of 20 Gy.

Exclusion Criteria:

* Pregnancy and lactating women.
* Cigarette smoker patients.
* Patients with severe comorbid illnesses or immunocompromised status.
* Patients receiving induction chemotherapy or those with previous head and neck radiotherapy. Patients using Amifostine during radiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-06-28 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Radiotherapy-Induced Oral Mucositis | From the start of radiotherapy to 2 weeks after the completion of radiotherapy.
  The incidence of any grade of oral mucositis will be measured in each group. This will be evaluated by recording the number of patients who develop oral mucositis during and after radiotherapy treatment.
Time to Onset of Oral Mucositis | From the start of radiotherapy to the onset of oral mucositis, monitored daily during radiotherapy and up to 2 weeks after completion of radiotherapy.
  The time from the start of radiotherapy to the onset of any grade of oral mucositis in groups I, II, III, and V (control group). This will be measured by tracking the number of days until the first appearance of mucositis symptoms.
Severity of Oral Mucositis | Assessed weekly during radiotherapy and up to 2 weeks after the completion of radiotherapy.
  The severity of oral mucositis will be measured using the World Health Organization (WHO) criteria for grading oral mucositis, which includes objective symptoms (redness, edema, wound development) and subjective symptoms (dysphagia, mucosal severity). Mucositis will be classified into grades:
  Grade 0: No change or erythema without pain. Grade 1: Pain with or without erythema, no ulcers. Grade 2: Oral erythema and ulcers, but the patient can eat solid and liquid food.
  Grade 3: Oral erythema and ulcers, the patient can eat only liquid/puree food. Grade 4: Severe oral ulcers; patient cannot eat solid or liquid food.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Aref, BDS, MS, Principal Investigator — Mansoura University
Locations (1):
- Mansoura university, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim HJ, Kang SU, Lee YS, Jang JY, Kang H, Kim CH. Protective Effects of N-Acetylcysteine against Radiation-Induced Oral Mucositis In Vitro and In Vivo. Cancer Res Treat. 2020 Oct;52(4):1019-1030. doi: 10.4143/crt.2020.012. Epub 2020 Jun 18. PMID 32599978